CLINICAL TRIAL: NCT00921817
Title: Validation of a Body Composition Method for Infants and Children
Brief Title: Body Composition in Infants and Children
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Aline Andres, PhD, University of Arkansas for Medical Sciences
Other Study IDs: 109498
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: healthy children

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — two urine samples are collected during the study visit
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will test a new method for measuring body fat and muscle in infants and children: QMR.

ELIGIBILITY:
Inclusion Criteria:

* healthy child
* weighing between 0 and 110 pounds

Exclusion Criteria:

* child has condition that may affect growth or bone development
* child has chronic disease
* child has disorder of carbohydrate metabolism
* child takes medication that could affect bone density
* child has any type of nonremovable metal

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: healthy children weighing between 0 and 110 pounds
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Body Composition | one-time visit

CONTACTS AND LOCATIONS:
Overall Officials: Aline Andres, PhD, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States